CLINICAL TRIAL: NCT04625842
Title: Quality Improvement Actions on the Radiotherapy Ward: Focus Group Interview Study on Patient Experiences and Satisfaction
Brief Title: Focus Group Interview Study on Patient Experiences and Satisfaction
Acronym: RT_Focus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has not been started since
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Mark De Ridder, Professor in oncology, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-087
Record Dates: First submitted 2020-03-05; First posted 2020-11-12 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Patient Satisfaction; Patient Preference
Keywords: Quality of care
MeSH Terms: conditions — Patient Satisfaction; Patient Preference

STUDY DESIGN:
Intervention Model Description: Focus group interview study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient focus group (Experimental): Patients who received radiation treatment
  Interventions: Other: Focus group interview
- Family focus group (Experimental): Family of patients who received radiation treatment
  Interventions: Other: Focus group interview

INTERVENTIONS:
Other: Focus group interview — Group interview with patients who received radiation treatment

SUMMARY:
In order to improve quality of care at the department, the investigators will perform a focus group interview study with patients and family members. They will perform 6 (3 in the French, and 3 in the Dutch language) focus group interviews with patients and 6 (3 in the French, and 3 in the Dutch language) with family members.

DETAILED DESCRIPTION:
In order to improve quality of care at the department, the investigators will perform a focus group interview study with patients and family members. They will perform 6 (3 in the French, and 3 in the Dutch language) focus group interviews with patients and 6 (3 in the French, and 3 in the Dutch language) with family members. Following research questions will be answered:

* What elements of care (ie infrastructure, interpersonal contact, information, communication) are good to the opinion of patients and family members?
* What elements of care can be improved?
* What are priorities in improvement of the care for patients and families?
* What actions could possibly be taken in order to improve the care for future patients?

Because the radiotherapy ward exists of 3 clusters, one per type of treatment conducted, the investigators will perform 6 focus group interviews with patients (3 in the French, and 3 in the Dutch language) and 6 focus group interviews with family members (3 in the French, and 3 in the Dutch language).

Investigators will collect sex, main diagnosis (of patients), age and nationality of all participants at the beginning of each focus group interview. They will transcribe all interviews verbatim and analyze them in Nvivo software as provided by the VUB. Participant characteristics will be analyzed by descriptive statistics.

ELIGIBILITY:
Inclusion criteria for patients:

* Patients (18+) who were treated for cancer, receiving radiotherapy, and followed thereafter in the UZ Brussel
* Dutch and French speaking
* Start date of treatment max 6 months before inclusion
* Estimated sample size: 5-8 x 6 patients

Inclusion criteria for family members:

* All family members (+18) of patients who were treated for cancer, receiving radiotherapy, and followed thereafter in the UZ Brussel
* Dutch and French speaking
* Start date of treatment of patient max 6 months before inclusion
* Estimated sample size: 5-8 x 6 family members

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of care | immediately after treatment
  To identify elements of care that need improvement by using open ended interview questions and interaction between different participants
Problem solving | immediately after treatment
  To identify solutions for problems in care by using open ended interview questions and interaction between different participants

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided